CLINICAL TRIAL: NCT07193524
Title: Assessment of the Feasibility of Using a Preoperative Surgical Fracture Analysis Tool
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Responsible Party: Principal Investigator, Derek S. Stenquist, MD, MD, Massachusetts General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2024P003282
Record Dates: First submitted 2025-09-24; First posted 2025-09-26 (Actual); Last update posted 2025-09-26 (Actual); Status verified 2025-09

CONDITIONS: Tibia Fractures; Trauma (Including Fractures); Surgical Planning
Keywords: 3D; Tibia fracture; Surgical Planning; Fracture Analysis
MeSH Terms: conditions — Wounds and Injuries; Tibial Fractures

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- 3D Analysis Group (Experimental)
  Interventions: Device: 3D Fracture Analysis Tool

INTERVENTIONS:
Device: 3D Fracture Analysis Tool — Based on a pre-operative computed tomography (CT) scan, fractured bone fragments of a proximal tibia are segmented and aligned to achieve adequate fracture reduction.
  Bone material properties for each fragment are derived from Hounsfield Units (HU) of the CT scan, based on internal density calibration with air, fat, muscle, and cortical bone. Screws and implants are then modelled based on the manufacturer's design and material properties Placement of off-the-shelf plate and screws can be analyzed and support a personalized plan on how to individually treat a patient with a specific fracture pattern and anatomical biometric data.
  Surgeons can define up to three approaches (different placement of implants and screws) to be visualized and analyzed for construct stability.
  The surgeons will receive a visualization of the fracture, fracture-reduction, implant and screw placement in 3D as well as a comparison of construct stabilites of the submitted approaches

SUMMARY:
This study aims to evaluate a preoperative fracture analysis tool that uses 3D visualization and biomechanical modeling to assist surgeons in planning screw and plate fixation for complex tibial plateau fractures. By simulating different fixation strategies based on patient-specific CT data, the tool provides insights into construct stability, potentially improving surgical precision and reducing intraoperative uncertainty. The study also investigates the tool's feasibility within current clinical workflows without altering the standard of care.

ELIGIBILITY:
Inclusion Criteria:

* Age above 18
* lower extremity fracture

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-09-10 (Actual); Primary Completion 2027-09 (Estimated); Study Completion 2028-09 (Estimated)

PRIMARY OUTCOMES:
Feasibility of incorporating the preoperative software plan based on surgeon's feedback | From enrollment to day after surgery
  Surgeons will fill out a questionnaire after the surgery to assess the clinical feasibility of the analysis tool.

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Massachusetts General Hospital, Boston, Massachusetts
  - Brigham and Women's Hospital, Boston, Massachusetts

IPD SHARING:
Plan to Share IPD: Yes
IPD used in the results publication.